CLINICAL TRIAL: NCT05182489
Title: Lumbar Fusion With Micro and Nano-textured Titanium Interbody Cages - A Single-Blinded Randomized Controlled Trial Evaluating Adaptix™ Versus PEEK Cages
Brief Title: Adaptix RCT Evaluating Adaptix™ Versus PEEK Cages
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Andrew Grossbach, Principal Investigator, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021H0244
Record Dates: First submitted 2021-12-09; First posted 2022-01-10 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Spinal Canal Stenosis; Spondylolisthesis; Osteophyte; Bony Growth Formation; Degenerative Disc Disease
MeSH Terms: conditions — Spinal Stenosis; Spondylolisthesis; Osteophyte; Intervertebral Disc Degeneration

STUDY DESIGN:
Intervention Model Description: All subjects will be randomized in the trial to receive either the Medtronic titanium or the PEEK cage supplemented with a pedicle screw system and milled local autograft bone supplemented with GRAFTON™ DBM DBF. Subject randomization will be stratified according to smoking status. Subjects will be blinded to their group status for the duration of the study assessments and procedures (24 months post-operatively).
Who Masked: Participant
Masking Description: Subjects will be blinded to their group status for the duration of the study assessments and procedures (24 months post-operatively).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Medtronic Adaptix™ titanium implants (Experimental): This arm will use Medtronic Adaptix™ titanium implants supplemented with a pedicle screw system. Both cages will be used in conjunction with a 50:50 mixture of autograft: allograft using milled local autograft bone and GRAFTON™ DBM DBF (no iliac crest autograft will be utilized).
  Interventions: Device: Medtronic Adaptix™ titanium implants
- Medtronic CAPSTONE® PEEK cage (Active Comparator): This arm will use Medtronic CAPSTONE® PEEK cage supplemented with a pedicle screw system. Both cages will be used in conjunction with a 50:50 mixture of autograft: allograft using milled local autograft bone and GRAFTON™ DBM DBF (no iliac crest autograft will be utilized).
  Interventions: Device: Medtronic CAPSTONE® PEEK cage

INTERVENTIONS:
Device: Medtronic Adaptix™ titanium implants — Patients who will be having a spinal fusion procedure as part of their standard of care treatment will be randomized to receive either the Medtronic titanium or the PEEK cage supplemented with a pedicle screw system and milled local autograft bone supplemented with GRAFTON DBM DBF. In order to assess fusion, patients will undergo a research-only CT Scan at 6 months post-surgery.
  Arms: Medtronic Adaptix™ titanium implants
Device: Medtronic CAPSTONE® PEEK cage — Medtronic CAPSTONE® PEEK cage
  Arms: Medtronic CAPSTONE® PEEK cage

SUMMARY:
The purpose of this randomized controlled trial is to assess and compare radiographic and clinical outcomes in patients who are to undergo combined interbody/posterolateral lumbar fusion procedures, supplemented with pedicle screw instrumentation, using one of the following interbody cages; the Medtronic Adaptix™ cage with roughened micro and nano-textured titanium surfaces or the CAPSTONE® poly-ether-ether-ketone cage.

DETAILED DESCRIPTION:
The randomized controlled trial will prospectively evaluate the efficacy of Medtronic Adaptix™ titanium implants supplemented with a pedicle screw system as compared to a Medtronic CAPSTONE® PEEK cage currently used in routine fashion for lumbar interbody fusion procedures. This study will capture clinical and radiographic outcomes on patients up to 2 years postoperatively. Both cages will be used in conjunction with a 50:50 mixture of autograft: allograft using milled local autograft bone and GRAFTON™ DBM DBF (no iliac crest autograft will be utilized).

This single-centered study will enroll up to 100 subjects, with subjects followed for 24 months post-surgery. All subjects enrolled in the study will be recruited from a pool of subjects eligible for combined interbody/posterolateral lumbar fusion surgery. The inclusion/exclusion criteria are listed below.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is scheduled to undergo combined interbody and posterolateral spinal fusion surgery using either the Medtronic Adaptix™ titanium cage or Medtronic CAPSTONE® PEEK cage in conjunction with a 50:50 mixture of local autograft and GRAFTON™ DBM DBF, and supplementation with a pedicle screw system.
2. Subject must be over the age of 18 years old.
3. Subject has been unresponsive to conservative care for a minimum of 6 months.
4. The subject must in the investigator's opinion, be psychosocially, mentally, and physically able to fully comply with this protocol including the required follow-up visits, the filling out of required forms, and have the ability to understand and give written informed consent.

Exclusion Criteria:

1. Subjects with previous lumbar arthrodesis surgery.
2. Subjects requiring additional bone grafting materials other than local autograft bone or GRAFTON™ DBM DBF.
3. Subject has inadequate tissue coverage over the operative site.
4. Subject has an open wound local to the operative area, or rapid joint disease, bone absorption, or osteoporosis.
5. Subject has a condition requiring medications that may interfere with bone or soft tissue healing (i.e., oral or parenteral glucocorticoids, immunosuppressives, methotrexate, etc.).
6. Subject has an active local or systemic infection.
7. Subject has a metal sensitivity/foreign body sensitivity.
8. Subject is allergic to antibiotics (gentamicin) or processing solutions found in GRAFTON™.
9. Subject is morbidly obese, defined as a body mass index (BMI) greater than 45.
10. Subject has any medical condition or extenuating circumstance that, in the opinion of the investigator, would preclude participation in the study.
11. Subject is currently involved in another investigational drug or device study that could confound study data.
12. Subject has a history (present or past) of substance abuse (recreational drugs, prescription drugs or alcohol) that in the investigator's opinion may interfere with protocol assessments and/or with the subject's ability to complete the protocol required follow-up.
13. Subjects who are pregnant or plan to become pregnant in the next 12 months or who are lactating.
14. Subject is involved in or planning to engage in litigation or receiving Worker's Compensation related to neck or back pain.
15. Subject is a prisoner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-11-19 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Fusion rate at 6 months | 6 months
  A subject will be considered a success if fusion is a Grade BSF-3 at 6 months. The primary outcome measure of effectiveness will be determined by the fusion rate at 6 months post-operatively in subjects implanted with either titanium cage as compared to the PEEK cage.

SECONDARY OUTCOMES:
Timing of fusion | 24 months
  Secondary measures of effectiveness will be determined by the principal investigator by evidence and timing of fusion observed in X-rays post-operatively (3, 6, 12, and 24 months).

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Wexner Medical Center Neurological Surgery, Columbus, Ohio, United States

REFERENCES:
- [Background] Anjarwalla NK, Brown LC, McGregor AH. The outcome of spinal decompression surgery 5 years on. Eur Spine J. 2007 Nov;16(11):1842-7. doi: 10.1007/s00586-007-0393-z. Epub 2007 May 23. PMID 17520297
- [Background] Banik BL, Riley TR, Platt CJ, Brown JL. Human Mesenchymal Stem Cell Morphology and Migration on Microtextured Titanium. Front Bioeng Biotechnol. 2016 May 10;4:41. doi: 10.3389/fbioe.2016.00041. eCollection 2016. PMID 27243001
- [Background] Fernyhough JC, Schimandle JJ, Weigel MC, Edwards CC, Levine AM. Chronic donor site pain complicating bone graft harvesting from the posterior iliac crest for spinal fusion. Spine (Phila Pa 1976). 1992 Dec;17(12):1474-80. doi: 10.1097/00007632-199212000-00006. PMID 1471005
- [Background] Gittens RA, Olivares-Navarrete R, McLachlan T, Cai Y, Hyzy SL, Schneider JM, Schwartz Z, Sandhage KH, Boyan BD. Differential responses of osteoblast lineage cells to nanotopographically-modified, microroughened titanium-aluminum-vanadium alloy surfaces. Biomaterials. 2012 Dec;33(35):8986-94. doi: 10.1016/j.biomaterials.2012.08.059. Epub 2012 Sep 16. PMID 22989383
- [Background] Hangai M, Kaneoka K, Kuno S, Hinotsu S, Sakane M, Mamizuka N, Sakai S, Ochiai N. Factors associated with lumbar intervertebral disc degeneration in the elderly. Spine J. 2008 Sep-Oct;8(5):732-40. doi: 10.1016/j.spinee.2007.07.392. Epub 2007 Nov 26. PMID 18037353
- [Background] Kurtz SM, Devine JN. PEEK biomaterials in trauma, orthopedic, and spinal implants. Biomaterials. 2007 Nov;28(32):4845-69. doi: 10.1016/j.biomaterials.2007.07.013. Epub 2007 Aug 7. PMID 17686513
- [Background] Laurencin C, Khan Y, El-Amin SF. Bone graft substitutes. Expert Rev Med Devices. 2006 Jan;3(1):49-57. doi: 10.1586/17434440.3.1.49. PMID 16359252
- [Background] Laurie SW, Kaban LB, Mulliken JB, Murray JE. Donor-site morbidity after harvesting rib and iliac bone. Plast Reconstr Surg. 1984 Jun;73(6):933-8. doi: 10.1097/00006534-198406000-00014. PMID 6374708
- [Background] Lee CS, Hwang CJ, Lee DH, Kim YT, Lee HS. Fusion rates of instrumented lumbar spinal arthrodesis according to surgical approach: a systematic review of randomized trials. Clin Orthop Surg. 2011 Mar;3(1):39-47. doi: 10.4055/cios.2011.3.1.39. Epub 2011 Feb 15. PMID 21369477
- [Background] Long EG, Buluk M, Gallagher MB, Schneider JM, Brown JL. Human mesenchymal stem cell morphology, migration, and differentiation on micro and nano-textured titanium. Bioact Mater. 2019 Sep 19;4:249-255. doi: 10.1016/j.bioactmat.2019.08.001. eCollection 2019 Dec. PMID 31667441
- [Background] Nemoto O, Asazuma T, Yato Y, Imabayashi H, Yasuoka H, Fujikawa A. Comparison of fusion rates following transforaminal lumbar interbody fusion using polyetheretherketone cages or titanium cages with transpedicular instrumentation. Eur Spine J. 2014 Oct;23(10):2150-5. doi: 10.1007/s00586-014-3466-9. Epub 2014 Jul 12. PMID 25015180
- [Background] Olivares-Navarrete R, Hyzy SL, Hutton DL, Erdman CP, Wieland M, Boyan BD, Schwartz Z. Direct and indirect effects of microstructured titanium substrates on the induction of mesenchymal stem cell differentiation towards the osteoblast lineage. Biomaterials. 2010 Apr;31(10):2728-35. doi: 10.1016/j.biomaterials.2009.12.029. Epub 2010 Jan 6. PMID 20053436
- [Background] Olivares-Navarrete R, Hyzy SL, Gittens RA 1st, Schneider JM, Haithcock DA, Ullrich PF, Slosar PJ, Schwartz Z, Boyan BD. Rough titanium alloys regulate osteoblast production of angiogenic factors. Spine J. 2013 Nov;13(11):1563-70. doi: 10.1016/j.spinee.2013.03.047. Epub 2013 May 14. PMID 23684238
- [Background] Quint U, Wilke HJ. Grading of degenerative disk disease and functional impairment: imaging versus patho-anatomical findings. Eur Spine J. 2008 Dec;17(12):1705-13. doi: 10.1007/s00586-008-0787-6. Epub 2008 Oct 7. PMID 18839226
- [Background] Santos ER, Goss DG, Morcom RK, Fraser RD. Radiologic assessment of interbody fusion using carbon fiber cages. Spine (Phila Pa 1976). 2003 May 15;28(10):997-1001. doi: 10.1097/01.BRS.0000061988.93175.74. PMID 12768137
- [Background] Summers BN, Eisenstein SM. Donor site pain from the ilium. A complication of lumbar spine fusion. J Bone Joint Surg Br. 1989 Aug;71(4):677-80. doi: 10.1302/0301-620X.71B4.2768321.
- [Background] Younger EM, Chapman MW. Morbidity at bone graft donor sites. J Orthop Trauma. 1989;3(3):192-5. doi: 10.1097/00005131-198909000-00002. PMID 2809818